CLINICAL TRIAL: NCT02008175
Title: Evaluation of Conventional Collagen Crosslinking in Young Keratoconus.
Brief Title: Conventional Collagen Crosslinking in Young Keratoconus
Acronym: PED-CXL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vasan Eye Care Hospital (Other)
Responsible Party: Principal Investigator, Dr.ANAND PARTHASARATHY, Dr. Ramesh Hariharan, Dr. Anand Parthasarathy, Vasan Eye Care Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PED_CXL
Record Dates: First submitted 2013-12-02; First posted 2013-12-11 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Keratoconus
Keywords: paediatric, keratoconus, collagen cross linking
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conventional CXL (Experimental): Crosslinking was done according to the standard protocol using hypo-osmolar riboflavin to saturate the cornea following epithelial debridement and ultra - violet light of 370nm with energy density of 3 milliwatts/sq.cm with riboflavin and distilled water alternated every 2 minutes was used for the procedure.
  Interventions: Radiation: Conventional CXL

INTERVENTIONS:
Radiation: Conventional CXL — Crosslinking was done according to the standard protocol using hypo-osmolar riboflavin (<0.1%) to saturate the cornea following epithelial debridement and ultra - violet light of 370nm with energy density of 3 milliwatts/cm2 with riboflavin and distilled water alternated every 2 minutes was used for the procedure..
  Other Names: Conventional collagen cross linking, C3R, Dresden protocol.

SUMMARY:
Keratoconus is a chronic progressive non - inflammatory disorder characterised by progressive steepening and thinning of cornea and high myopic astigmatism, accounting for poor visual acuity in such individuals. Keratoconus seems to be more advanced on presentation, in young patients.

The investigators intend to evaluate the effectiveness of conventional collagen cross linking in young patients diagnosed with keratoconus.

DETAILED DESCRIPTION:
Keratoconus is progressive ectatic corneal disorder characterised by progressive corneal thinning, steep corneal curvatures and usually associated with high irregular myopic astigmatism.

The major problems concerning keratoconus in young patients are;

1. Rapid rates of progression in young keratoconic corneas as compared to adults.
2. Poor biomechanical properties of young corneas.
3. Poor quality of vision, which predisposes to a very poor quality of life.
4. High rates of complications and failure post keratoplasty in young patients.

The investigators intend to evaluate the effectiveness of conventional collagen crosslinking in young patients with keratoconus with regards to keratometric indices and visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and below.
* Patients diagnosed to have keratoconus at presentation and willing for follow - up at regular intervals post treatment.

Exclusion Criteria:

* Any disease causing abnormal topography other than keratoconus.
* Any ocular condition predisposing towards poor vision (retinal , lens problems)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Keratometric indices | 1 months
  The keratometric readings in the steepest and flattest meridians, along with the average K readings were compared pre and post treatment using conventional collagen cross linking technique at 1 month post cross linking.

SECONDARY OUTCOMES:
Improvement in vision | 12 months
  Comparison of visual rehabilitation was done as improvements noted in Snellen line numbers and best corrected visual acuity (B.C.V.A) converted to decimals, pre and post treatment at 1,3,6,12 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Anand Parthasarathy, Principal Investigator — Vasan Eye Care Hospital
Locations (1):
- Vasan Eye Care Hospital, Chennai, Tamil Nadu, India

REFERENCES:
- [Background] Vinciguerra P, Albe E, Frueh BE, Trazza S, Epstein D. Two-year corneal cross-linking results in patients younger than 18 years with documented progressive keratoconus. Am J Ophthalmol. 2012 Sep;154(3):520-6. doi: 10.1016/j.ajo.2012.03.020. Epub 2012 May 24. PMID 22633357
- [Background] Chatzis N, Hafezi F. Progression of keratoconus and efficacy of pediatric [corrected] corneal collagen cross-linking in children and adolescents. J Refract Surg. 2012 Nov;28(11):753-8. doi: 10.3928/1081597X-20121011-01. PMID 23347367
- [Background] Caporossi A, Mazzotta C, Baiocchi S, Caporossi T, Denaro R, Balestrazzi A. Riboflavin-UVA-induced corneal collagen cross-linking in pediatric patients. Cornea. 2012 Mar;31(3):227-31. doi: 10.1097/ico.0b013e31822159f6. PMID 22420024